CLINICAL TRIAL: NCT03889080
Title: Central Pain Location in SCN9A-associated SFN, an fMRI Pilot Study.
Brief Title: fMRI-study in Patients With Small Fiber Neuropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Ziekenhuis Maastricht (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Catharina G. Faber, Prof. Dr. C.G. Faber, Academisch Ziekenhuis Maastricht
Other Study IDs: fMRI-SFN
Record Dates: First submitted 2018-11-21; First posted 2019-03-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Small Fiber Neuropathy
Keywords: functional MRI; fMRI; pain
MeSH Terms: conditions — Small Fiber Neuropathy; Pain | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SCN9A-group: Patients with SCN9A-associated small fiber neuropathy
  Interventions: Diagnostic Test: functional MRI
- Skin biopsy: Patients with SFN confirmed with a decreased intra-epidermal nerve fiber density (IENFD)
  Interventions: Diagnostic Test: functional MRI
- Control: Age- and gender-matched healthy controls
  Interventions: Diagnostic Test: functional MRI

INTERVENTIONS:
Diagnostic Test: functional MRI — functional MRI scan of the brain

SUMMARY:
Small fiber neuropathy (SFN) is a form of peripheral neuropathy, which is characterized by neuropathic pain and autonomic dysfunction. Mutations in SCN9A, the gene encoding for the voltage-gated sodium channel NaV1.7, are associated with SFN. SCN9A-associated SFN often results in chronic neuropathic pain, which is difficult to treat. Chronic neuropathic pain may cause structural and functional changes in the brain. Until now, only one small study examined the structural and functional changes of the brain in SFN patients. No studies have been performed in strictly defined SFN patients.

Therefore, it would be interesting to explore whether in SFN patients with an SCN9A mutation, the genotype will lead to a distinct brain activation pattern on functional MRI (fMRI) and if the integrity or structural connectivity of the brain is altered using diffusion tensor imaging (DTI). This may provide a better understanding of the pathophysiological pathways for chronic pain and might serve as a biomarker for evaluating therapy.

The objective of this study is to explore whether there is an indication whether patients with SCN9A-associated SFN have an abnormal brain activation pattern on resting state fMRI and during advanced thermal stimulation and altered structural connectivity on DTI versus SFN patients without a mutation and versus age- and gender-matched healthy controls. With this knowledge, objective pain measurement for patients with SFN may serve as a biomarker in evaluating efficacy of targeted therapy.

DETAILED DESCRIPTION:
Small fiber neuropathy (SFN) is a form of peripheral neuropathy, which is characterized by neuropathic pain and autonomic dysfunction. It is caused by dysfunction of the Aδ-fibers and C-fibers. SFN is diagnosed if typical SFN symptoms are present, in combination with an additional abnormal skin biopsy and/or abnormal quantitative sensory testing. The minimal prevalence of SFN is estimated to be 53/100.000. SFN has a comprehensive list of causes. The etiology encompasses metabolic, toxic, auto immune, infectious, and hereditable causes. Mutations in SCN9A, the gene encoding for the voltage-gated sodium channel NaV1.7, are associated with SFN, and can be found in 10-15% of SFN patients. The symptomatic treatment of SFN is generally disappointing. Until now, antidepressants and anticonvulsants are mostly recommended for SFN with limited pain reduction, often leading to chronic daily pain experience. Understanding the pathophysiology of pain and identifying plausible specific pain genotype-phenotype relations, might lead to improved treatment strategies. Therefore, the focus should extend beyond the scope of peripheral mechanisms of the nervous system and should include searching for pain complex central, thus brain based, mechanisms and patterns (a pain network of somatosensory, limbic and associate structures).

The International Association for the Study of Pain defined pain as 'an unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage'. A painful stimulus activates the peripheral nociceptors and is transmitted through the small fibers, via the dorsal horn in the spinal cord, to the brain. Pain stimuli are processed in the cortex, subcortical structures, and the midbrain. In the cortical area the somatosensory, anterior cingulate, prefrontal, and insular cortex are the most important structures, whereas important subcortical areas encompass the hippocampus, basal ganglia, amygdala, and thalamus. Furthermore, the cerebellum is suggested as an important area contributing to pain sensation.

Chronic pain may lead to structural changes in the brain, and imaging revealed morphological alterations in gray matter (both an increase and a decrease). The pattern of alterations may differ among different pain syndromes and may be reversible.

Functional imaging studies have displayed specific brain activity patterns in patients with different types of pain syndromes. Recently, also in a small SFN patients study functional connectivity changes using a 3.0 Tesla scanner were shown. However, whether a specific activation pattern can be seen depends on many factors, such as type of brain imaging modality.7 It is conceivable that a particular type of pain (stimulus) may enhance a specific pain brain pattern, but also specific person factors (for example gender and genetic factors) may influence the pain activation network. Psychological modulation as well as chronicity of pain may influence the activation network, and should therefore be taken into account. Furthermore the specific location of pain can display different kinds of patterns because of partially somatotopic organization, such as described in the S1 cortex. To date, in human no functional imaging studies using a 7.0 Tesla fMRI-scan have been performed.

Until now, an objective tool to measure pain is lacking. Most studies in pain syndromes including patients with SFN have been using a great variety of surrogate pain scales, such as the Visual Analogue Pain Scale (VAS), the Pain Intensity Numerical Rating Scale, the Brief Pain Inventory and the Neuropathic pain scale (NPS). Therefore, an objective measure for pain would be a great advantage.

In this study, patients with a SCN9A-associated SFN will be analyzed to determine possible central nervous system pain network patterns. The voltage-gated sodium channel NaV1.7 plays a central role in pain processing. Research in rats revealed areas of the brain that express Nav1.7 channels. These channels were restricted to the hypothalamic/preoptic area, brain stem, and the subfornical organ. Our goal is to examine whether gain-of-function mutations in NaV1.7 may lead to a specific pain pattern in the human brain by scanning with a 3.0 Tesla fMRI-scan. Some patients will be included to undergo an extra fMRI-brain scan (Tesla 7.0). Due to the high field strength, new opportunities have arisen for brain imaging. The newly acquired ultra high resolution facilitates the possibility of more detailed anatomical imaging. When the 7.0 Tesla fMRI-scan appears to yield more useful information than the 3.0 Tesla fMRI-scan, the first-mentioned will be used for follow-up studies.

The aim of this study is to determine the resting state and the effect on heat stimuli of patients with SCN9A-associated SFN on fMRI and the changes in structural connectivity using diffusion tensor imaging (DTI). This may provide a better understanding of the pathophysiological pathways for chronic pain. If successful, fMRI/DTI might be an additional tool as biomarker for evaluating therapy, and may contribute in the evaluation of novel therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

Patient group (SCN9A-associated SFN)

* Male and/or female subjects between the ages of 18 and 80 years.
* Presence of a clinical diagnosis of SFN, according to international criteria, and presence of confirmed abnormality on intra-epidermal nerve fiber density evaluation (IENFD) and/or Quantitative Sensory Testing (QST).
* A mutation in the SCN9A gene, confirmed by sequencing, with possible, probable or certain pathogenicity according to international criteria.
* Presence of pain due to SFN for at least 3 months and an average self-reported pain score of at least 5.
* Subjects must give informed consent by signing and dating an informed consent form.

Patient group (SFN without a gene mutation):

* Male and/or female subjects between the ages of 18 and 80 years.
* Presence of a clinical diagnosis of SFN, according to international criteria, including a decreased intra-epidermal nerve fiber density IENFD in skin biopsy.
* No mutation in the SCN9A, SCN10A or SCN11A gene, confirmed by sequencing.
* Presence of pain due to SFN for at least 3 months and an average self-reported pain score of at least 5.
* Subjects must give informed consent by signing and dating an informed consent form.

Control group

* Male and/or female subjects between the ages of 18 and 80 years.
* Subjects must give informed consent by signing and dating an informed consent form

Exclusion Criteria:

For all groups:

* Major depression according to DSM-V criteria or a history of major psychiatric disease.
* (History of) alcohol abuse
* HADS ≥ 14
* Subjects who have another pain syndrome than small fiber neuropathy.
* Contraindications for undergoing MRI: pacemaker, metallic foreign body (including aneurysm clip in the brain), claustrophobia, pregnancy, neurostimulator, pacemaker or other kinds of implanted devices or insulin pump. In case of cardiac valve replacement of ossicular replacement prosthesis the radiologist will be consulted.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients can only participate when they are living in the Netherlands.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-10-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
BOLD during heat stimulation | Once (1 day)
  BOLD (blood-oxygen-level dependent) signal in 3 study cohorts (individuals with SCN9A mutation with small fiber neuropathy, individual with SCN9A mutation without small fiber neuropathy and matched, healthy controls) during heat stimulation. [ Time Frame: 1 day, single timepoint] Difference in BOLD signal measured by functional magnetic resonance imaging (fMRI) between study cohorts in primary somatosensory cortex, thalamus, dorsal striatum and ventral striatum.
BOLD during cold stimulations | Once (1 day)
  BOLD (blood-oxygen-level dependent) signal in 3 study cohorts (individuals with SCN9A mutation with small fiber neuropathy, individual with SCN9A mutation without small fiber neuropathy and matched, healthy controls) during cold stimulation. [ Time Frame: 1 day, single timepoint] Difference in BOLD signal measured by functional magnetic resonance imaging (fMRI) between study cohorts in primary somatosensory cortex, thalamus, dorsal striatum, and ventral striatum.

SECONDARY OUTCOMES:
Resting state | Once (1 day)
  Resting state functional connectivity signal in 3 study cohorts (individuals with SCN9A mutation with small fiber neuropathy, individual with SCN9A mutation without small fiber neuropathy and matched, healthy controls) [Time Frame: 1 day, single timepoint]
  Difference in resting-state functional connectivity strength measured by functional magnetic resonance imaging (fMRI) between study cohorts in default-mode, sensorimotor and salience networks.
Fractional anisotropy | Once (1 day)
  Fractional anisotropy in 3 study cohorts (individuals with SCN9A mutation with small fiber neuropathy, individual with SCN9A mutation without small fiber neuropathy and matched, healthy controls) [Time Frame: 1 day, single timepoint]
  Difference in fractional anisotropy measured by diffusion tensor imaging and tract based spatial statistics between study cohorts. Whole brain analysis will be performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Gool R, Far A, Drenthen GS, Jansen JFA, Goijen CP, Backes WH, Linden DEJ, Merkies ISJ, Faber CG, Upadhyay J, Hoeijmakers JGJ. Peripheral Pain Captured Centrally: Altered Brain Morphology on MRI in Small Fiber Neuropathy Patients With and Without an SCN9A Gene Variant. J Pain. 2024 Mar;25(3):730-741. doi: 10.1016/j.jpain.2023.10.002. Epub 2023 Nov 3. PMID 37921732